CLINICAL TRIAL: NCT03067727
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled Phase III Trial Investigating the Efficacy and Safety of FE 999901 Vaginal Insert in Pregnant Women at Term (41 Weeks of Gestation) Requiring Cervical Ripening
Brief Title: A Randomised Trial Investigating the Efficacy and Safety of a Vaginal Insert in Pregnant Women at Term
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000262
Record Dates: First submitted 2017-02-09; First posted 2017-03-01 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2018-09

CONDITIONS: Cervical Ripening
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dinoprostone vaginal insert (Experimental)
  Interventions: Drug: Dinoprostone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dinoprostone — The DVI contains 10 mg Dinoprostone
  Other Names: CERVIDIL®; PROPESS®
  Arms: Dinoprostone vaginal insert
Drug: Placebo — The placebo product is identical with the active product except that it does not contain Dinoprostone.
  Arms: Placebo

SUMMARY:
To demonstrate the efficacy of dinoprostone vaginal insert (DVI) for cervical ripening success (either bishop score (BS) ≥7 or vaginal delivery) within 12 hours of vaginal insert administration

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at term (≥ 41 weeks 0 day and ≤ 41 weeks 6 days of gestation) at the Baseline visit
* Candidate for pharmacologic induction of labour
* Singleton pregnancy with live infant in vertex presentation
* Baseline BS ≤ 4 at the Baseline visit
* Parity ≤ 3 (parity is defined as one or more births live or stillbirths after 22 weeks 0 day gestation)
* Written informed consent

Exclusion Criteria:

* Women in labour
* Presence of uterine or cervical scar including scar from previous caesarean section, and previous cone biopsy of the cervix and loop electrosurgical excision procedure (LEEP)
* Uterine abnormality e.g. bicornuate uterus
* Administration of oxytocin, any cervical ripening or labour inducing agents (including mechanical methods) or a tocolytic drug within 7 days prior to IMP administration. Magnesium sulfate is permitted if prescribed as treatment for preeclampsia or pregnancy induced hypertension
* Presence of the following conditions/symptoms:

Systolic blood pressure > 160 mmHg or diastolic blood pressure > 110 mmHg. Platelets < 100,000/µL. Increased liver function tests (2x upper limits of normal range). Severe, persistent right upper quadrant/epigastric pain. Progressive renal insufficiency: Creatinine > 1.1 mg/dL, Doubling of creatinine in the absence of other renal disease. Pulmonary edema. New onset cerebral or visual disturbances

* Suspected or confirmed cephalopelvic disproportion and/or fetal malpresentation
* Diagnosed congenital abnormalities, not including polydactyly
* Suspected or confirmed intrauterine growth retardation (≤ 1.5 SD of mean normal estimated fetal weight for dates)
* Any evidence of fetal compromise at baseline visit (e.g., non-reassuring fetal heart rate pattern, meconium staining, history of non-reassuring fetal status or abnormal umbilical artery Doppler wave form)
* Intake of medication with aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) at baseline visit
* Ruptured membranes
* Suspected clinical chorioamnionitis
* Current pelvic inflammatory disease, unless adequate prior treatment has been instituted
* Fever (axillary temperature ≥ 38.0 °C) at the Baseline visit
* Any condition in which vaginal delivery is contraindicated (eg., placenta previa or any unexplained vaginal bleeding at any time after 24 weeks 0 day during this pregnancy)
* Known or suspected allergy to, dinoprostone other prostaglandins or any constituent of IMP
* Any condition urgently requiring delivery
* History of asthma or glaucoma
* Unable to comply with the protocol
* Any other medical condition which in the judgement of the investigator would impair participation in the trial

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
The proportion of women with cervical ripening success | Within 12 hours of vaginal insert administration
  Defined as either Bishop Score (BS) ≥7 or a vaginal delivery

SECONDARY OUTCOMES:
Proportion of nulliparous and multiparous subjects with cervical ripening success | Within 12 hours of Investigational Medicinal Product (IMP) administration
  Collected labour data and delivery data
Proportion of subjects delivering vaginally | Within 12 hours of IMP administration
  Collected labour and delivery data
Proportion of subjects delivering vaginally | Within the first admission to hospital
  Collected labour data and delivery data
Proportion of subjects with a BS increase ≥3 points from baseline | Within 12 hours of IMP administration
  Measured by BS assessments
Proportion of subjects who have a caesarean delivery within the first admission to hospital | At time of delivery
  Data collected during the first admission to hospital
Proportion of subjects who receive pre-delivery oxytocic drugs and dose of pre-delivery oxytocic drugs | From the IMP removal to delivery
  Collected pre-delivery data
Proportion of subjects who undergo mechanical cervical ripening | At least 60 minutes after the removal of the IMP
  Collected labour data
Duration of mechanical cervical ripening for subjects who undergo mechanical Cervical ripening | Time from at least 60 minutes after the removal of the IMP until end of any mechanical ripening
  Measured as start date and time of first mechanical ripening and the end date and time of last mechanical ripening
Proportion of subjects with BS ≥7 | At onset of labour
  Among those having onset of labour while IMP is in-situ
Time from IMP administration to onset of active labour | Interval from IMP administration to onset of active labour
  Within the first admission to hospital
Time from IMP administration to vaginal delivery, caesarean delivery and any delivery | Interval from IMP administration to delivery
  Within the first admission to hospital
Type, frequency and intensity of intrapartum adverse events (AEs), postpartum AEs and neonatal AEs | From obtaining the informed consent through end of trial (expected average of up to 1 week)
  Assessed up to time when the subjects are discharged from the hospital
Type, frequency and intensity of intrapartum AEs | From onset of labour to the removal of the IMP
  Assessed up to time when the deliveries occur
Change in maternal parameters of vital signs (blood pressure, heart rate and body temperature) | From baseline through end of trial (expected average of up to 1 week)
  Assessed up to time when the subjects are discharged from the hospital
Change in maternal parameters of haematology, clinical chemistry and urinalysis | From baseline to end of trial (expected average of up to 1 week)
  Assessed up to time when the subjects are discharged from the hospital
Proportion of neonates with Apgar Score <7 | 5 minutes post-birth
  Measured as Apgar Score assessments
pH in umbilical artery blood samples | At birth
  pH evaluation
Rate of admission to neonatal intensive care unit (NICU) for at least 24 hours | After delivery
  Admission/discharge data from NICU

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (20):
- Japan (20):
  - Osaka Medical Center and Research Institute for Maternal and Child Health, Izumi, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Itabashi Chuo Medical Center, tabashi City, Tokyo
  - Asahi General Hospital, Chiba
  - University of Tsukuba Hospital, Ibaraki
  - Hori Hospital, Kanagawa
  - Aizenbashi Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Rinku General Medical Center, Osaka
  - Juntendo University Hospital, Tokyo
  - Keio University Hospital, Tokyo
  - Seibo Hospital, Tokyo
  - Showa University Hospital, Tokyo
  - St.Luke's International Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Tokyo
  - Tokyo Metropolitan Tama Medical Center, Tokyo
  - Keiyu Hospital, Yokohama

REFERENCES:
- [Result] Itoh H, Ishii K, Shigeta N, Itakura A, Hamada H, Nagamatsu T, Ishida T, Bungyoku Y, Falahati A, Tomisaka M, Kitamura M. Efficacy and safety of controlled-release dinoprostone vaginal delivery system (PROPESS) in Japanese pregnant women requiring cervical ripening: Results from a multicenter, randomized, double-blind, placebo-controlled phase III study. J Obstet Gynaecol Res. 2021 Jan;47(1):216-225. doi: 10.1111/jog.14472. Epub 2020 Oct 22. PMID 33094550